CLINICAL TRIAL: NCT00474409
Title: A Multicenter, Placebo-Controlled, Double-Blind Study To Evaluate The Efficacy And Safety Of Betahistine Mesilate In The Treatment Of Patients With Vertigo Caused By Cerebral Infarction In Posterior Circulation
Brief Title: A Study To Evaluate The Efficacy And Safety Of Betahistine Mesilate In The Treatment Of Patients With Vertigo Caused By Cerebral Infarction In Posterior Circulation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to poor enrollment, this study was withdrawn/ terminated.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRS-CHN-001
Record Dates: First submitted 2007-05-03; First posted 2007-05-16 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Vertigo
Keywords: Vertigo; Posterior circulation infarction
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Merislon

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Betahistine Mesilate in the treatment of patients with vertigo caused by Cerebral Infarction in posterior circulation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have a clinical diagnosis of posterior circulation infarction and vertigo occurring within 1 month after the infarction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Changes in the European Evaluation of Vertigo (EEV) scale in 4 weeks. | 4 weeks

SECONDARY OUTCOMES:
The duration of the vertigo symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yong Jun, Principal Investigator — Beijing Tiantan Hospital
Locations (4):
- China (4):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Shanghai Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality